CLINICAL TRIAL: NCT07005518
Title: Study of the Relationship Between Curarization and Pneumoperitoneum in Laparoscopic Surgery
Acronym: PneumandTOF
Status: Not yet recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PneumandTOF
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Laparoscopic Surgery; Neuromuscular Blocking Agents; Pneumoperitoneum
Keywords: pneumoperitoneum pressure; curarization
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the group will be composed of patients undergoing laparoscopic surgery: the group will be made up of patients undergoing laparoscopic surgery and willing to take part in the pressure monitoring study.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This is a non-interventional observational study. It will simply look at the data and compare them between the monitors provided.

SUMMARY:
The number of surgical procedures is increasing worldwide (1). Laparoscopic surgery is one of the surgical techniques that has become indispensable. Laparoscopic surgery is less invasive than laparotomy. Laparoscopic surgery is performed in several stages, one of which involves the creation of a peritoneal detachment. This detachment is achieved by the addition of a gas (CO2), which requires total relaxation of the abdominal muscle fibers. To achieve this, it is advisable to administer a muscle relaxant called curare (2). Curare-induced neuromuscular block, its depth and its release must be monitored during surgery. Curares act as acetylcholine antagonists, inducing neuromuscular block by competing with this neurotransmitter. In France, only one type of device, called an accelerometer, is used to monitor curarization. This device couples electrical stimulation of a nerve with an accelerometer. Curarization can be said to be deep, moderate, residual or absent. Despite curarization appearing deep to the accelerometer, operating conditions do not always seem ideal for abdominal contraction. Indeed, the muscles tested with this device do not concern the muscles involved in laparoscopic surgery.

A currently unexploited surgical parameter, variation in insufflation pressure, could change our approach to intraoperative curarization.

DETAILED DESCRIPTION:
Curarization is a fundamental part of surgical management. The administration of these drugs enables intubation and facilitates surgical work. However, these molecules need to be monitored at every stage, from anesthetic induction to patient awakening. Today, a single device is used in operating theatres to monitor the depth of patient curarization. This tool is used on a daily basis, and its use is strongly recommended by the various learned societies associated with anesthesia. Its use in operating theatres is compulsory by law. The device is used either on the ulnar nerve, generating a contraction of the adductor muscle of the thumb, or on the facial nerve, generating a contraction of the orbicularis muscle of the eye. This reflects the curarization of the laryngeal and diaphragmatic muscles. The device delivers repetitive electrical stimulation to these nerves, producing a muscle contraction. The number of muscle contractions in response to these stimulations, and the strength developed by the fourth response compared with the first, indicates the depth of curarization. These measurements are called a train of four.

While performing a train-of-four on the thumb adductor produces measured, quantifiable data, this is absolutely not the case for the orbicularis of the eye, which provides only crude, unreliable data intraoperatively.

Laparoscopic surgery, on the other hand, is a minimally invasive technique that has become increasingly popular in recent decades. It requires deep intraoperative curarization.

This surgical technique can be used for a wide range of urological, visceral and gynecological procedures.

During laparoscopic surgery, insufflation pressure is delivered via trocars into the patient's abdominal cavity. This pressure comes from a column supplied via a carbon dioxide (CO2) cylinder. Initially, a pressure is generated and adjusted at the surgeon's request (3). This pressure creates a space known as the pneumoperitoneum. In the event of insufficient pneumoperitoneum to enable surgery to be performed under optimum conditions, potentially due to a lack of deep curarization, the insufflation pressure is increased at the surgeon's request. This surgical technique is nonetheless prone to causing significant projected pain. As Madsen's study (4) suggests, lowering the insufflation pressure could therefore result in less pain.

By hypothesizing that imperfect curarization would lead to contraction of the abdominal muscles, generating intra-abdominal overpressure. This study investigates the role of intra-abdominal pressure variation in laparoscopic surgery and its correlation with the accelerometer used in current practice. If this hypothesis proves to be true, the expected benefits would be improved operating conditions for surgeons, reduced intra-operative risks of perforation and organ damage, and improved patient comfort in the post-operative period.

ELIGIBILITY:
Major patient, operated on by robot-assisted laparoscopic surgery, by two surgeons targeted for their similar working surgical technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-inclusion criteria: patients whose anesthetic maintenance is performed with Propofol IACP, patients who have undergone more than 3 intra-abdominal surgical procedures, patients with conversion to laparotomy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure | one day
  Evaluate the relationship between variation in intra-abdominal pressure and depth of curarization.

SECONDARY OUTCOMES:
secondary outcome | 3 month
  Study whether there is a link between variation in abdominal pressure level and postoperative pain.
secondary outcome | one day
  To study whether taking insufflation pressure into account reduces the need for intraoperative curare administration.
secondary outcome | one day
  To study whether taking into account variations in insufflation pressure can reduce the dose of curare administered.

IPD SHARING:
Plan to Share IPD: Undecided